CLINICAL TRIAL: NCT04196517
Title: Can the Patient Activated Learning System (PALS) Serve as a Better Model for Nutrition Education Than Other Online-based Educational Material?
Brief Title: PALS for Nutrition Education
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 paused study temporarily due to no clinical encounters
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-11021133
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Nutrition Disorders
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - PALS (Experimental): The Patient Activated Learning System (Palsforhealth.com)
  Interventions: Other: Educational Tool, PALS
- Arm 2 - WebMD (Experimental): WebMD.com
  Interventions: Other: WebMD

INTERVENTIONS:
Other: Educational Tool, PALS — The Patient Activated Learning System is a free, health education platform.
  Arms: Arm 1 - PALS
Other: WebMD — WebMD is a widely used educational platform for health information.
  Arms: Arm 2 - WebMD

SUMMARY:
The overall goal of this inquiry is to determine whether PALS is more effective than comparable online resources at educating patients in the outpatient clinic setting about nutrition. Participants will be randomly assigned to view either a PALS article or WebMD article on the same nutrition topic. Participants will then fill out a post-survey to assess knowledge uptake and attitudes regarding healthy eating.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age.
* Ability to speak and read in English.
* Passing the screener - Mini-Mental Status Examination.
* Patient at WCIMA clinic on Upper East Side of Manhattan, NY.

Exclusion Criteria:

* Non-English speakers
* Inability to read in English
* Being younger than 18
* Not passing the screener
* Not a patient at WCIMA clinic on Upper East Side of Manhattan, NY.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Knowledge, as measured by assessment questions on the nutrition information provided | Day 1, Immediately after reading article

SECONDARY OUTCOMES:
E-health usability, as measured by questions from the Kelly et al. scale | Day 1, Immediately after reading article
  Questions to understand the user's understanding, preference and trust of the information based on a 5-point likert scale with 5 being strongly agree in favor.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Safford, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No